CLINICAL TRIAL: NCT04628026
Title: A Randomized, Placebo-Controlled Phase III Study of Induction and Consolidation Chemotherapy With Venetoclax in Adult Patients With Newly Diagnosed Acute Myeloid Leukemia or Myelodysplastic Syndrome With Excess Blasts-2
Brief Title: Phase III Study of Induction and Consolidation Chemotherapy With Venetoclax in Patients With Newly Diagnosed AML or MDS-EB-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Doehner, Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMLSG31-19/HO501/AbbVieB18-982
Record Dates: First submitted 2020-11-03; First posted 2020-11-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: adult patients
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind with open label dose-finding run-in part
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): standard chemotherapy in combination with venetoclax
  Interventions: Drug: Venetoclax; Combination Product: Standard chemotherapy; Other: Allogeneic stem cell transplantation
- 2 (Placebo Comparator): standard chemotherapy in combination with placebo
  Interventions: Drug: Placebo; Combination Product: Standard chemotherapy; Other: Allogeneic stem cell transplantation

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be administered in Induction cycle 1, Induction cycle 2 and in the chemo consolidation therapy in addition to the standard chemotherapy
  Arms: 1
Drug: Placebo — Placebo will be administered in Induction cycle 1, Induction cycle 2 and in the chemo consolidation therapy in addition to the standard chemotherapy
  Arms: 2
Combination Product: Standard chemotherapy — Induction cycle 1: Patients will receive cytarabine 200 mg/m2 continuous IV (days 1-7) and daunorubicin 60 mg/m2 IV (days 1-3). Induction cycle 2: Patients ≤ 60 yrs will receive cytarabine 1000 mg/m2 BID (3h IV), days 1-4, and daunorubicin 60 mg/m2 IV (days 1-3). Patients >60 yrs will receive cytarabine 1000 mg/m2 BID (3h IV), days 1-4 without daunorubicin.
  Consolidation chemotherapy with intermediate doses of cytarabine. Patients ≤60 yrs will receive up to 3 cycles of IDAC (single dose 1500 mg/m2 every 12 hours, days 1-3). Patients who are >60 yrs will receive up to 3 cycles of IDAC with single doses of 1000 mg/m2, every 12 hours, days 1-3. In patients >60 yrs less than 3 cycles of IDAC or dose-reduced IDAC (500 mg/m2 per single dose) may be given based on an individual risk assessment.
Other: Allogeneic stem cell transplantation — Generally, patients will proceed to allogeneic HCT upon completion of remission induction chemotherapy. It is however allowed, as per investigator's discretion, for a patient to receive 'bridging' consolidation chemotherapy in exceptional cases of delay towards transplantation. At baseline, HLA-compatible donor search must be initiated as soon as possible, first among siblings and second in the world donor bank for unrelated donors or cord blood. In order to avoid inappropriate delay in cases where no suitable sibling is present, high-resolution HLA typing should be performed immediately after registration, enabling a more rapid matched-unrelated donor search. In case no sibling or unrelated donor can be identified, haploidentical allogeneic HCT is allowed. Conditioning and GVHD prophylaxis will take place according to institutional guidelines. Patients who undergo allogeneic HCT will not receive venetoclax during conditioning, engraftment or after hematologic recovery.

SUMMARY:
A Randomized, Placebo-Controlled Phase III Study of Induction and Consolidation Chemotherapy With Venetoclax in Adult Patients With Newly Diagnosed Acute Myeloid Leukemia or Myelodysplastic Syndrome With Excess Blasts-2

DETAILED DESCRIPTION:
Prospective, multicenter, double-blind, randomized, placebo-controlled phase 3 clinical study. The randomized phase of the study will be preceded by a feasibility run-in dose-escalation phase in patients with AML in which the venetoclax dose for the phase 3 part will be established.

After the feasibility run-in phase, eligible patients will be randomized to intensive chemotherapy with venetoclax or placebo. Patients will receive two cycles of induction chemotherapy; patients achieving CR or CRi after two cycles will continue with consolidation treatment according to initial randomization, and according to Cooperative Group-specific consolidation regimens or investigator choice. Patients achieving morphologic leukemia-free state (MLFS) only, may also continue consolidation treatment on protocol. Assignment to either allogeneic hematopoietic cell transplantation (HCT), conventional chemotherapy or autologous HCT will be done according to institutional standards, and based on (prognostic) disease characteristics, individual patient assessment, and established comorbidity risk scores (e.g., HCT-CI score).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed acute myeloid leukemia (AML) according to the International Consensus Classification (ICC).
2. Age ≥ 18 and ≤ 75 years.
3. Patients considered eligible for intensive chemotherapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Molecular analysis centrally performed in AMLSG and HOVON laboratories.
6. Adequate renal function as evidenced by serum creatinine ≤ 2.0 × upper limit of norm (ULN) or creatinine clearance >40 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR).
7. Adequate hepatic function as evidenced by:

   * Serum total bilirubin ≤ 2.5 × ULN unless considered due to Gilbert's disease, or leukemic involvement following approval by the Principal Investigators or Trial Coordinators of the study
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3.0 × ULN, unless considered due to leukemic involvement following approval by the Principal Investigators or Trial Coordinators.
8. No prior chemotherapy for AML, except hydroxyurea for up to 14 days during the diagnostic screening phase for the control of peripheral leukemic blasts in patients with leukocytosis (e.g., white blood cell [WBC] counts > 25x109/L); patients may have had previous treatment with erythroid stimulating agents (ESA) or hypomethylating agents (HMAs) for an antecedent phase of MDS; ESA and HMAs have to be stopped at least four weeks before start of study treatment.
9. Patients must not have received a known strong or moderate CYP3A inducer 7 days before start of study treatment. Patients must have no known medical conditions requiring chronic therapy with moderate or strong CYP3A inducers.
10. Female patient must either:

    * Be of nonchildbearing potential:

      * Postmenopausal (defined as at least 1 year without any menses)
      * Documented surgically sterile (e.g. documented hysterectomy, bilateral oophorectomy, bilateral salpingectomy or congenital sterile) or status post hysterectomy (at least 1 month prior to screening)
    * Or, if of childbearing potential (not surgically sterile and not postmenopausal)

      * Not planning to become pregnant during the study and for 6 months after the final study drug administration
      * And have a negative urine or serum pregnancy test at screening
      * And, if heterosexually active, agree to consistently apply one highly effective* method of birth control in combination to a barrier method for the duration of the study and for 27 weeks after the final study drug administration

        *Highly effective forms of birth control include
      * Consistent and correct usage of established hormonal contraceptives that inhibit ovulation for at least 1 month prior to taking study drug. (hormonal contraception is only a highly effective method of birth control, if a combined [estrogen and progestogen containing] hormonal contraception or a progestogen-only hormonal contraception - both associated with inhibition of ovulation - is used.
      * Established intrauterine device (IUD) or intrauterine system (IUS)
      * Bilateral tubal occlusion
      * Vasectomy - a vasectomy is highly effective contraception method provided the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.
      * Male is sterile due to a bilateral orchiectomy.
      * Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual activity during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient.

        *List is not all inclusive. Prior to enrolment, the investigator is responsible for confirming patient will utilize highly effective forms of birth control in combination with a barrier method according to locally accepted standards during the protocol defined period.
      * Female patient must agree not to breastfeed starting at screening and throughout the study period, and for 2 months and 1 week after the final study drug administration.
      * Female patient must not donate ova starting at screening and throughout the study period, and for 27 weeks after the final study drug administration.
11. Men must use a latex condom during any sexual contact with WOCBP, even if they have undergone a successful vasectomy and must agree to avoid to father a child (while on therapy and for 27 weeks after the final study drug administration). In addition, their female partners of childbearing potential have to use a highly effective method of birth control.
12. Male patient must not donate sperm starting at screening and throughout the study period and for 27 weeks after the final study drug administration.
13. Able to understand and willing to sign an informed consent form (ICF).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | 6 months/16 months after inclusion of last patient
  EFS in adult patients with newly diagnosed AML, defined as the time from randomization to treatment failure, death from any cause, or relapse after achieving CR or CRi, or start of new therapy due to confirmed molecular relapse whichever occurs first. Treatment failure is defined as not attaining CR or CRi after induction chemotherapy, and EFS event time for treatment failure is Day 1 of post-randomization
Frequency of dose-limiting toxicities (DLTs) during the observation period (Primary safety endpoint during dose-finding phase) | after cycle 1 (maximal day 42)
  Frequency of dose-limiting toxicities (DLTs) during the observation period (from start of cycle 1 up to a maximum of day 42, or until the start of cycle 2)

SECONDARY OUTCOMES:
Overall Survival (OS) | 6 months/16 months/28 months after inclusion of last patient
  OS in patients with newly diagnosed AML
CR/CRi rate | 2 months
  Complete remission (CR/CRi) rate in newly diagnosed AML patients defined as the proportion of AML patients with CR/CRi after induction chemotherapy
CR rate | 2 months
  Complete remission (CR) rates in newly diagnosed AML patients defined as the proportion of AML patients with CR after induction chemotherapy
Event Free Survival (EFS) including CRh | 6 months/16 months after inclusion of last patient
  EFS in adult patients with newly diagnosed AML, defined as the time from randomization to treatment failure, death from any cause, or relapse after achieving CR, CRh or CRi, or start of new therapy due to confirmed molecular relapse whichever occurs first. Treatment failure is defined as not attaining CR, CRh or CRi by end of induction chemotherapy, i.e. if a patient's best response during or at completion of the induction treatment is less than CR/CRh/CRi
Rates of complete remission without measurable residual disease (CRMRD-) after induction therapy | 2 months
  Rates of complete remission without measurable residual disease (CRMRD-) after induction therapy, defined as the proportion of AML patients achieving CR with negativity for a genetic marker by RT-qPCR, and/or with negativity by multi-color flow cytometry, if studied pre-treatment
Relapse-free survival (RFS) in newly diagnosed AML patients | 16 months after inclusion of last patient
  Relapse-free survival (RFS) in newly diagnosed AML patients, defined as the time from achievement of a remission (CR/CRh/CRi) following curative therapy (induction and consolidation), to relapse, or start of new therapy due to confirmed molecular relapse or death from any cause
Cumulative incidence of relapse (CIR) in newly diagnosed AML patients | 16 months after inclusion of last patient
  Cumulative incidence of relapse (CIR) in newly diagnosed AML patients
Cumulative incidence of death (CID) | 16 months after inclusion of last patient
  Cumulative incidence of death (CID) in newly diagnosed AML patients.
EQ-5D-5L questionnaire of the EuroQoL (EQ) group, among AML patients | at study entry, 2 months, 3 months, 6 months
  Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated using a 5 level (5L) scale from 1 (minimum) to 5 (maximum). Higher score values mean a worse outcome.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) among AML patients | at study entry, 2 months, 3 months, 6 months
  All sub scales and single items have values from 1 (minimum) to 100 (maximum) points. A higher point value represents a better condition in terms of the functional scales and quality of life. In the symptomal sub scales a higher point value represents a worse condition.
Patient Reported Outcome Measurement Information System (PROMIS) Cancer Fatigue short form among AML patients | at study entry, 2 months, 3 months, 6 months
  The 7-item PROMIS Cancer Fatigue Short Form assesses the frequency of fatigue in the past seven days (7). Table 2 presents a list of the items. Items are measured on a five point scale (1 = never; 5 = always) and summed, after reverse scoring item 7, with higher scores indicating greater fatigue (worse condition).
CR/CRh rate | 2 months
  Complete remission (CR/CRh) rate in newly diagnosed AML patients defined as the proportion of AML patients with CR/CRh after induction chemotherapy
Rates of complete remission without measurable residual disease (CR/CRh MRD-) after induction therapy | 2 months
  Rates of complete remission without measurable residual disease (CR/CRh MRD-) after induction therapy, defined as the proportion of AML patients achieving CR/CRh with negativity for a genetic marker by RT-qPCR, and/or with negativity by multi-color flow cytometry, if studied pre-treatment
Rates of complete remission without measurable residual disease (CR/CRi MRD-) after induction therapy | 2 months
  Rates of complete remission without measurable residual disease (CR/CRi MRD-) after induction therapy, defined as the proportion of AML patients achieving CR/CRi with negativity for a genetic marker by RT-qPCR, and/or with negativity by multi-color flow cytometry, if studied pre-treatment

OTHER OUTCOMES:
Rates of CR+CRi in newly diagnosed AML patients after induction 1 | 1 month
  Rates of CR+CRi in newly diagnosed AML patients defined as proportion of AML patients achieving CR/CRi after first course of induction
Rates of CR in newly diagnosed AML patients after induction 1 | 1 month
  Rates of CR in newly diagnosed AML patients defined as proportion of AML patients achieving CR after first course of induction
EFS in newly diagnosed AML patients across different patient subgroups | 6 months/16 months after inclusion of last patient
  EFS in newly diagnosed AML patients across different groups are defined based on prognostic characteristics including age at randomization , risk category according to ELN 2022 recommendations, as well as specific AML genotypes
OS in newly diagnosed AML patients across different patient subgroups | 6 months/16 months/28 months after inclusion of last patient
  OS in newly diagnosed AML patients across different groups are defined based on prognostic characteristics including age at randomization , risk category according to ELN 2022 recommendations, as well as specific AML genotypes
CR/CRi rates in newly diagnosed AML patients across different patient subgroups | 2 months
  CR/CRi rates in newly diagnosed AML patients across different groups are defined based on prognostic characteristics including age at randomization , risk category according to ELN 2022 recommendations, as well as specific AML genotypes
CR rates in newly diagnosed AML patients across different patient subgroups | 2 months
  CR rates in newly diagnosed AML patients across different groups are defined based on prognostic characteristics including age at randomization , risk category according to ELN 2022 recommendations, as well as specific AML genotypes
RFS in newly diagnosed AML patients across different patient subgroups | 16 months after inclusion of last patient
  RFS in newly diagnosed AML patients across different groups are defined based on prognostic characteristics including age at randomization , risk category according to ELN 2022 recommendations, as well as specific AML genotypes
CIR in newly diagnosed AML patients across different patient subgroups | 16 months after inclusion of last patient
  CIR in newly diagnosed AML patients across different groups are defined based on prognostic characteristics including age at randomization , risk category according to ELN 2022 recommendations, as well as specific AML genotypes
CID in newly diagnosed AML patients across different patient subgroups | 16 months after inclusion of last patient
  CID in newly diagnosed AML patients across different groups are defined based on prognostic characteristics including age at randomization , risk category according to ELN 2022 recommendations, as well as specific AML genotypes
Frequency and severity of AE | 6 months
  Frequency and severity of AE according to CTCAE version 5.0 in newly diagnosed AML patients
Times to hematopoietic recovery | 6 months
  Times to hematopoietic recovery (absolute neutrophil counts ≥0.5 and ≥1.0 x 109/L; platelets ≥50 and ≥100 x 109/L) after each chemotherapy treatment cycle, defined as the time from the start of the cycle until recovery among AML patients
EFS with modified definition | 6 months/16 months after inclusion of last patient
  To evaluate the impact of venetoclax on EFS in newly diagnosed AML patients using modified endpoint definitions:
  o Modified EFS includes treatment failure defined as not achieving CR by end of induction chemotherapy assessed by investigator. The date of treatment failure is date of randomization. Patients achieving CRh or CRi are counted as events.
RFS with modified definition | 16 months after inclusion of last patient
  To evaluate the impact of venetoclax on RFS in newly diagnosed AML patients using modified endpoint definitions:
  o Modified RFS includes only subjects achieving CR
Rates of CR/CRh in newly diagnosed AML patients after induction 1 | 1 month
  Rates of CR/CRh in newly diagnosed AML patients defined as proportion of AML patients achieving CR/CRh after first course of induction
CR/CRh rates in newly diagnosed AML patients across different patient subgroups | 2 months
  CR/CRh rates in newly diagnosed AML patients across different groups are defined based on prognostic characteristics including age at randomization , risk category according to ELN 2022 recommendations, as well as specific AML genotypes

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Doehner, MD, Principal Investigator — University of Ulm
Locations (91):
- Austria (6):
  - Tirol Kliniken GmbH, Innsbruck
  - Kepler Universitaetsklinikum GmbH, Linz
  - Ordensklinikum Linz GmbH, Linz
  - Landeskrankenhaus (LKH) Rankweil, Interne E am Landeskrankenhaus Rankweil, Rankweil
  - Gemeinnuetzige Salzburger Landeskliniken Betriebsgesellschaft mbH, Salzburg
  - Hanusch Krankenhaus Der Wiener Gebietskrankenkasse, Vienna
- Belgium (6):
  - Ziekenhuis Aan De Stroom, Antwerp
  - Az St-Jan Brugge-Oostende A.V., Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Katholieke Universiteit te Leuven, Leuven
  - Algemeen Ziekenhuis Delta, Roeselare
  - CHU UCL NAMUR - Mont Godinne, Yvoir
- Estonia (2):
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Finland (2):
  - Helsinki University Central Hospital Meilahden Kolmiosairaala, Helsinki
  - Tampere University Hospital, Tampere
- Germany (50):
  - Klinikum Aschaffenburg-Alzenau gGmbH, Aschaffenburg
  - HELIOS Klinikum Bad Saarow GmbH, Bad Saarow
  - Charité Berlin - Campus Mitte, Berlin
  - Charité Berlin - Campus Benjamin Franklin, Berlin
  - Charité Berlin - Campus Virchow Klinikum, Berlin
  - Vivantes am Urban, Berlin
  - Vivantes Neukölln, Berlin
  - Vivantes Spandau, Berlin
  - Knappschaftskrankenhaus Bochum-Langendreer, Bochum
  - Uniklinikum Bonn, Bonn
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - Gesundheit Nord gGmbH Klinikverbund Bremen, Bremen
  - Klinikum Darmstadt GmbH, Darmstadt
  - St. Johannes Hospital Dortmund, Dortmund
  - Marien Hospital Duesseldorf GmbH, Düsseldorf
  - Klinikum Frankfurt Hoechst GmbH, Frankfurt
  - Justus-Liebig-Universitaet Giessen, Giessen
  - Wilhelm-Anton-Hospital Goch, Goch
  - Universitätsmedizin Greifswald, Greifswald
  - Univeritätsklinikum, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Asklepios Klinik St Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - KRH Klinikum Siloah, Hanover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Marien Hospital Herne, Herne
  - Universitaetsklinikum des Saarlandes AöR, Homburg
  - Wespfalz-Klinikum, Kaiserslautern
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - UNIVERSITÄTSKLINIKUM Schleswig-Holstein, Lübeck
  - Otto Von Guericke Universitaet Magdeburg, Magdeburg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, Mainz
  - Klinikum Hochsauerland GmbH, Meschede
  - Muhlenkreiskliniken AöR, Minden
  - Klinikum rechts der Isar der TU Muenchen AöR, München
  - Ortenauklinikum, Offenburg
  - Klinikum Oldenburg AöR, Oldenburg
  - Universitaetsklinikum Regensburg AöR, Regensburg
  - Universitaetsklinikum, Rostock
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Klinikum Traunstein, Traunstein
  - Barmherzige Brueder Trier gGmbH, Trier
  - Klinikum Mutterhaus der Borromaerinnen, Trier
  - Uniklinikum Tübingen, Tübingen
  - University Hospital Ulm, Ulm
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - Helios Universitaetsklinikum Wuppertal, Wuppertal
- Vilnius University Hospital Santaros Klinik, Vilnius, Lithuania
- Netherlands (20):
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - Meander Medisch Centrum, Amersfoort
  - Amsterdam UMC Stichting, Amsterdam
  - OLVG, Amsterdam
  - Rijnstate Ziekenhuis Stichting, Arnhem
  - Amphia Hospital, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Maxima Medisch Centrum, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - UMCG, Groningen
  - Medisch Centrum Leeuwarden B.V., Leeuwarden
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Maastricht University Medical Center+ (MUMC+), Maastricht
  - Sint Antonius Ziekenhuis Stichting, Nieuwegein
  - Radboudumc, Nijmegen
  - Erasmus MC - Daniel, Rotterdam
  - Hagaziekenhuis, locatie Leyweg, The Hague
  - UMCU, Utrecht
  - Isala Klinieken Stichting, Zwolle
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Stavanger Univ. Hosp.-Rogaland Hosp., Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olavs Hospital, Trondheim